CLINICAL TRIAL: NCT00751036
Title: Randomized Phase III Trial Comparing Nilotinib 800mg to Imatinib 800 mg for the Treatment of Patients With Advanced and/or Metastatic Gastrointestinal Stromal Tumors Refractory to Imatinib 400 mg
Brief Title: Nilotinib 800 Mg And Imatinib 800 Mg For The Treatment Of Patients With Gastrointestinal Stromal Tumors (Gist) Refractory To Imatinib 400 Mg
Acronym: MACS0375
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DBR01; 2010-019806-18
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nilotinib (Experimental): Patients who were assigned to this treatment group received 400 mg. nilotinib bid.
  Interventions: Drug: Nilotinib
- Imatinib (Active Comparator): Patients who were assigned to this treatment group received 400 mg. imatinib bid.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib hard gel capsules were supplied to the Investigators at dose strengths of 200 mg. Nilotinib is a novel agent, which has been approved for the treatment of chronic phase and accelerated phase Philadelphia-chromosome-positive CML in adult patients resistant to or intolerant to prior therapy that included imatinib.
  Other Names: Tasigna
  Arms: Nilotinib
Drug: Imatinib — Imatinib tablets were supplied at 100 mg and/or 400 mg dose strength. Imatinib is an approved agent for GIST. Efficacy of imatinib at a dose of 400 mg bid has been established in the setting of disease progression after the use of the conventional dose (400 mg qd).
  Arms: Imatinib

SUMMARY:
The study will investigate the comparative efficacy and safety of two oral inhibitors of Kit and PDGFR: nilotinib 400 mg bid, a novel agent, and imatinib 400 mg bid, an approved agent with an established efficacy.

DETAILED DESCRIPTION:
This is an international, randomized, open-label, double-arm, phase III trial that will be conducted in centers in Latin America, Asia, Europe and Canada. The study will be sponsored by Novartis Pharmaceuticals Corporation. Patient enrollment will be competitive and will have a duration of up to 30 months. An interim analysis is planned to occur when approximately 60% of the PFS events occurs. A total of 150 patients per arm will be enrolled in the study. Eligible patients will have advanced/metastatic, inoperable GIST of any anatomical location or recurrent GIST while on or post imatinib adjuvant therapy, with documented disease progression on therapy with imatinib 400 mg q.d.

ELIGIBILITY:
Inclusion Criteria:

* Provide a written informed consent.
* Male or female patients ≥ 18 years of age.
* Histologically confirmed diagnosis of GIST of any anatomical location, which is unresectable and/ or metastatic or recurrent.
* Documented disease progression according to RECIST 1.0. Documentation of progression required by either 2 CT scans or 2 MRI scans within 6 months prior to randomization (one image will document the lesion and the other will document the progression by lesion(s) growth or the presence of new lesion(s)). The interval between the 2 images should be no greater than 6 months apart. Scans will be provided to the selected imaging CRO.
* Documented disease progression must occur while on imatinib 400 mg PO q.d. Imatinib therapy could be for (1) unresectable GIST; (2) metastatic GIST; or (3) recurrent GIST while on imatinib adjuvant therapy or recurrent GIST post adjuvant imatinib therapy.
* Positive immunohistochemical staining for c-KIT (CD117) or negative staining for KIT, but with either positive staining for DOG1 or an identified mutation on KIT or PDGFR genes.
* Presence of at least one measurable lesion according to RECIST 1.0, defined as a lesion that can be accurately measured in at least one dimension (longest diameter) as ≥ 20 mm with conventional techniques (conventional CT or MRI scan) or as ≥ 10 mm with spiral CT scan. Lesions in previously irradiated areas can be considered measurable only if they have demonstrated clear evidence of progression since the radiotherapy.
* A performance status of 0, 1 or 2 according to the Eastern Cooperative Oncology Group (ECOG) scale (Oken et al 1982)(Appendix A).
* Adequate organ function, as indicated by all of the following:
* White blood cell (WBC) count ≥ 3500/mm3;
* Absolute neutrophil count (ANC) ≥1500/mm3;
* Hemoglobin ≥ 9.0 g/dL;
* Platelet count ≥ 100 x 109/L;
* Total bilirubin ≤ 1.5 X ULN (< 3.0 X ULN if related to disease);
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the ULN, unless liver metastases present, in which case AST and ALT have to be ≤ 5 times the ULN;
* Serum creatinine ≤ 1.5 times the ULN;
* Serum amylase and lipase ≤1.5 X ULN;
* Alkaline phosphatase ≤2.5 X ULN (≤ 5.0 X ULN if related to disease);
* Serum potassium, phosphorus, magnesium and calcium ≥ LLN [lower limit of normality] or correctable with supplements prior to first dose of study drug. (Total calcium corrected for serum albumin)
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration.
* Fertile patients (female) must agree to use an acceptable method of contraception to avoid pregnancy for the duration of the study and for 3 months after study termination.

Exclusion Criteria:

* Prior use of imatinib doses higher than 400 mg q.d. or prior use of any other tyrosine-kinase inhibitor.
* Tumor progression after stopping imatinib 400 mg q.d.
* No investigational cytotoxic drug ≤ 4 weeks (6 weeks for nitrosurea or mitomycin C) prior to the Screening Visit (V100) is allowed with the exception of imatinib therapy.
* Cytotoxic, or antineoplastic treatments, such as chemotherapy, immunotherapy, biological response modifiers, or radiotherapy.
* If the only measurable lesion was previously irradiated and has not shown clear evidence of progression since the radiotherapy, the patient cannot be included.
* Serious uncontrolled concomitant medical or psychiatric illness.
* Impaired cardiac function including any one of the following:
* LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) confirmed by ECHO or Muga
* Inability to determine the QT interval on ECG
* Complete left bundle branch block
* Right bundle branch block plus left anterior or posterior hemiblock
* Use of a ventricular-paced pacemaker
* Congenital long QT syndrome or a known family history of long QT syndrome
* History of or presence of clinically significant ventricular or atrial tachyarrhythmias
* Clinically significant resting bradycardia (<50 bpm);
* QTcF >450 msec on screening ECG (using the QTcF formula). If QTc >450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc;
* History or clinical signs of myocardial infarction within 1 year of study entry
* History of unstable angina within 1 year of study entry
* Other clinically significant heart disease (e.g., congestive heart failureor uncontrolled hypertension).
* Treatment with strong CYP3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. (Appendix B).
* Treatment with strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbitol, St John's Wort), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Patients using medication that have been documented to prolong QT interval (see Appendix B for complete list).
* Grade 3 or higher impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome).
* History of acute pancreatitis within one year of study entry or medical history of chronic pancreatitis.
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients with any other clinically significant medical or surgical condition which, according to investigators' discretion, should preclude participation; (i.e.: severe renal disease unrelated to tumor, active or chronic liver disease- hepatitis B or C virus carriers with normal liver function tests, as described above, can be included). This includes patient with an acquired bleeding disorder unrelated to cancer.
* Use of any investigational agent within 28 days prior to enrollment in the study or foreseen use of an investigational agent during the study.
* History of non-compliance to medical regimens or inability to grant consent.
* Women who are pregnant, breast feeding, or of childbearing potential without a negative serum pregnancy test at baseline. Male or female patients of childbearing potential unwilling to use effective barrier contraceptives throughout the trial and for 3 months following discontinuation of study drug. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Inability to comply with the study protocol.
* Patients with a history of CNS metastasis. Note: Patients without clinical signs and symptoms of CNS involvement are not required to have CT/MRI of the brain.
* Major surgery within 4 weeks prior to randomization or those who have not recovered from prior surgery

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
- Brazil (8):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Divinópolis, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- China (4):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- South Korea (3):
  - Novartis Investigative Site, Hwasun-gun, Jeollanam-do
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- Novartis Investigative Site, Caracas, Distrito Federal, Venezuela

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib | Imatinib
Started | 48 (Started = Treated) | 46 (Started = Treated)
Completed | 0 (Reason Not Completed = Reason for End of Treatment) | 0 (Reason Not Completed = Reason for End of Treatment)
Not Completed | 48 | 46
Not completed — Disease Progression | 28 | 29
Not completed — Adverse Event | 6 | 4
Not completed — Administrative Problems | 3 | 4
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Missing end of Treatment Page | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | Imatinib | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Customized [Number; unit: Participants]
  <65 years | 38 | 35 | 73
  ≥ 65 years | 9 | 11 | 20
  Missing | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is the time from date of randomization to the date of first documented progression or death due to any cause. If a participant has not had an event, progression-free survival is censored at the time of last adequate tumor assessment. Progression is defined according to modified RECIST criteria as at least a 20% increase in the sum of the longest diameter of target lesions, worsening of the non-target lesions or the appearance of one or more new lesions.
Time Frame: 24 months
Population: Full Analysis Set (FAS) consisted of all randomized patients. Following the intent to treat principle, patients were analyzed according to the treatment which they were assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 48 | 46
Days | 111.00 [83.00 to 190.00] | 120.00 [59.00 to 173.00]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: The Disease Control Rate (Complete Response(CR), Partial Response (PD) and Stable Disease (SD) rates for each treatment arm will be computed using the exact Clopper-Pearson interval estimation methodology. DCR is defined as the percentage of patients with a best overall response of • CR, i.e. at least two determinations of CR at least 4 weeks apart without loss of response between the determinations, • PR, i.e. at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) and without loss of PR between the determinations, or • SD lasting at least 24 weeks, i.e. at least one SD or better response at least 24 weeks after randomization (and not qualifying for CR or PR).
Time Frame: every 2 months until 24 months (end of study)
Population: Full analysis set (FAS): consisted of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment to which they were assigned at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 48 | 46
Percentage of Patients
  Disease Control Rate (CR, PR, or SD) | 54.2 [39.2 to 68.6] | 47.8 [32.9 to 63.1]
  Complete Response (CR) | 2.1 [0.1 to 11.1] | 0 [0 to 7.7]
  Partial Response (PR) | 4.2 [0.5 to 14.3] | 6.5 [1.4 to 17.9]
  Stable Disease (SD) | 47.9 [33.3 to 62.8] | 41.3 [27.0 to 56.8]
  Progressive Disease (PD) | 25.0 [13.6 to 39.6] | 37.0 [23.2 to 52.5]
  Unknown (UNK) | 20.8 [NA to NA] — Confidence Interval was not assessed for Unknown. | 15.2 [NA to NA] — Confidence Interval was not assessed for Unknown.

3. Secondary Outcome: Time to Treatment Failure
Description: TTF, defined as the time from date of randomization to the earliest of date of the first objective tumor progression, date of death due to any cause, or date of discontinuation due to reasons other than 'Protocol deviation' or 'Administrative problems'.
Time Frame: Time from date of radomization to the earliest date of the first objective tumor, death or discontinuation, assesed until 24 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 48 | 46
Days | 90.00 [56.00 to 166.00] | 112.00 [58.00 to 171.00]

4. Secondary Outcome: Overall Survival (OS)
Description: . OS is defined as the time from the date of randomization to the date of death due to any cause or the date of last contact prior to or on the date of data cutoff. The median time to overall survival and its associated 95 % CI will be derived, for each treatment arm, using the time to event analysis based on Kaplan-Meier methodology.
Time Frame: time from the date of randomization to the date of death due to any cause or the date of last contact prior to or on the date of data cutoff, assesed until 24 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 48 | 46
Days | 737 [342.00 to NA] — Study was terminated early. | 594.00 [357.00 to NA] — Study was terminated early.

ADVERSE EVENTS:
Groups:
- Nilotinib 800 mg: Patients who were assigned to this treatment group received 400 mg. nilotinib bid.
- Imatinib 800 mg: Patients who were assigned to this treatment group received 400 mg. imatinib bid.
Arm/Group | Nilotinib 800 mg | Imatinib 800 mg
Serious Adverse Events (participants affected / at risk) | 12/48 | 10/46
Other Adverse Events (participants affected / at risk) | 39/48 | 41/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib 800 mg (N=48) | Imatinib 800 mg (N=46)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 2 | 1
Drug ineffective (General disorders) | 1 | 1
Performance status decreased (General disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tumour excision (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib 800 mg (N=48) | Imatinib 800 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 14 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Eyelid oedema (Eye disorders) | 0 | 6
Abdominal distension (Gastrointestinal disorders) | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Ascites (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 14
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 12 | 20
Vomiting (Gastrointestinal disorders) | 10 | 13
Asthenia (General disorders) | 6 | 5
Face oedema (General disorders) | 0 | 9
Fatigue (General disorders) | 10 | 12
Oedema peripheral (General disorders) | 3 | 9
Pyrexia (General disorders) | 8 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 0
Influenza (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 8 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 1
Blood albumin decreased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 8 | 0
Blood calcium decreased (Investigations) | 0 | 3
Blood potassium decreased (Investigations) | 1 | 6
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Neutrophil count decreased (Investigations) | 2 | 4
White blood cell count decreased (Investigations) | 2 | 8
Decreased appetite (Metabolism and nutrition disorders) | 6 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 8 | 2
Dysuria (Renal and urinary disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 2
Hypertension (Vascular disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Patients were limited (planned 300, Actual 94). Early termination of study; not sufficient power to test the original primary hypothesis with respect to PFS. Only descriptive analyses were carried out for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.